CLINICAL TRIAL: NCT06310707
Title: A Randomized Controlled Study to Identify Clinically Actionable Arrhythmia Using the ePatch® Extended Wear Holter vs. Standard Wear Holter
Brief Title: Arrhythmia Identification in Syncope Patients: ePatch® Versus 24h Holter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. Slow Enrollment. 2. Issues regarding reimbursement of product
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EU RCT: ePatch vs 24h Holter; 2022-A02338-35 (Other: ANSM, French competent authority); EA4/071/23 (Other: German Ethics Committee_Charité Universitätsmedizin Berlin)
Record Dates: First submitted 2023-11-29; First posted 2024-03-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Arrythmia; Syncope
Keywords: Clinically Actionable Arrhythmia; Symptoms of syncope
MeSH Terms: conditions — Arrhythmias, Cardiac; Syncope

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized, unblinded, two-arm study, to include approximately 128 subjects treated with the ePatch Extended Wear Holter (worn for 7 days) and approximately 128 subjects treated with a Standard Wear Holter (worn for 24 hours). Randomization will be balanced for gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ePatch® Extended Wear Holter (EWH) Arm (Experimental): Participants will undergo long-term continuous ambulatory ECG recording of 7-day duration
  Interventions: Device: ePatch ® Extended Wear Holter (EWH)
- Standard of Care (No Intervention): Participants will undergo 24 hours of continuous ECG recording.

INTERVENTIONS:
Device: ePatch ® Extended Wear Holter (EWH) — Diagnostic Test: Extended ECG investigation
  • An ambulatory ECG recordings with a duration of 7 days using Philips ePatch (https://www.myheartmonitor.com/device/epatch/) will be applied
  Arms: ePatch® Extended Wear Holter (EWH) Arm

SUMMARY:
This study is a Multi-center, prospective, randomized, unblinded, two-arm study to assess if 7-days of cardiac monitoring using the ePatch Holter results in identification of more clinically actionable arrythmia for patients with symptoms of syncope than standard 24 hour Holter monitoring.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized, unblinded, two-arm study to assess if 7-days of cardiac monitoring using the ePatch Holter results in identification of more clinically actionable arrythmia for patients with symptoms of syncope than standard 24 hour Holter monitoring. Approximately 256 adult subjects with symptoms of syncope will be randomized 1:1 to wear either the Philips ePatch Extended Wear Holter (7 day) or Standard Wear Holter (24 hours). Randomization will be balanced for gender.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Recommended for ambulatory cardiac Holter monitoring due to symptoms of syncope
3. Able to comply with continuous ECG monitoring for up to 7 days
4. Able and willing to replace the Patch electrode at home
5. Capable of providing voluntary informed consent and mentally and physically willing and able to be compliant with the protocol, including the follow-up visit(s)

Exclusion Criteria:

1. Patient with chronic Atrial Fibrillation (AF)
2. Patient with implanted pacemaker/defibrillator
3. Patient with known allergy to adhesive materials and/or hydrogel
4. Patient with broken, damaged, or irritated skin where ECG patch will be placed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield (frequency) of clinically actionable arrythmia | Up to 7 days
  In patients indicated for cardiac monitoring due to syncope, show that the diagnostic yield (frequency) of clinically actionable arrythmia with 7 days of monitoring using the ePatch Extended Wear Holter is superior to what would be seen with the Standard Wear Holter (24 hours).

SECONDARY OUTCOMES:
Number of Atrial Fibrillation (AF) diagnoses > 30 seconds | Up to 7 days
  Number of Atrial Fibrillation (AF) diagnoses > 30 seconds with 7 days of monitoring using the ePatch Extended Wear Holter vs. Standard Wear Holter (24 hours).
Occurrence of symptomatic events | Up to 7 days
  Occurrence of symptomatic events in 7 days of monitoring using the ePatch Extended Wear Holter vs. Standard Wear Holter (24 hours).
Number of Clinically actionable arrhythmia | Up to 7 days
  Clinically actionable arrhythmia yield vs days of data collected
  * Analysis for all patients
  * Analysis for patients with sporadic symptoms (less than one per day)
Patient Quality of Life as measured by EQ-5D-5L | Up to 7 days
  Patient Quality of Life will be measured using the EQ-5D-5L at 24-hours (Standard Wear Holter and ePatch) and at end of service (ePatch arm only, at 7 days). The EQ-5D-5L stands for EuroQol, 5 dimensions, 5 levels.
  EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). Higher scores mean a worse outcome.
Patient Quality of Life as measured by Patient Experience Survey | Up to 7 days
  Patient Quality of Life will be measured using survey data at 24-hours (Standard Wear Holter and ePatch) and at end of service (7 days for ePatch arm)
  Each question in the Patient Experience Survey has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). Higher scores mean a worse outcome.
Cost related to cardiac monitoring | Up to 7 days
  - Compare clinical workflow costs from 7 days of cardiac monitoring using the ePatch Extended Wear Holter vs. 24 hours of cardiac monitoring with Standard Wear Holter.
Time Holter is worn/ removed | Up to 7 days
  Compare time Holter is worn/removed
  - Assess via diary

CONTACTS AND LOCATIONS:
Locations (2):
- Hospices Civils de Lyon - Hôpital Cardiologique Louis Pradel, Bron, France
- Deutsches Herzzentrum der Charité (DHZC) - Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No